CLINICAL TRIAL: NCT03473938
Title: Adjustable Balloons for Weight Loss: A Higher Yield of Responders Compared With Non-Adjustable Balloons
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: Clínica Opcíon Médica Barcelona (Unknown); Optimal Clinic Tel Aviv (Unknown); University of Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-IK-Intragastric-Balloon
Record Dates: First submitted 2018-03-14; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Intragastric balloons; Adjustable gastric balloon; Weight loss plateau; Intolerance
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spatz3 AIGB: Patients with implanted Spatz3 AIGB balloon.
  Interventions: Device: Spatz3 AIGB

INTERVENTIONS:
Device: Spatz3 AIGB — Implantation of Spatz3 AIGB balloon.

SUMMARY:
Intragastric balloon degree of efficacy and duration of effect can be variable and unpredictable. The Spatz Adjustable intragastric balloon (AIGB) was developed to extend implantation to 1 year, decrease balloon volume for intolerance and increase volume for diminishing effect. The aim of the study was to determine the utility/efficacy and responder rate with the Spatz3 AIGB.

DETAILED DESCRIPTION:
The results of the Spatz adjustable balloon system have been reported in four studies with weight losses of 24.4 kg (48.8% excess weight loss - EWL), 21.6 kg (45.7% EWL),17.2 kg (42.9% EWL) and 16.3 kg (67.4% EWL), respectively. The responder rate (>25% EWL) was 88.5% in one recent study.

The authors report and analyze the results of 227 Spatz3 patients retrospectively reviewed in 3 centers- some adjusted and some not adjusted during the course of their 1-year implantation - to determine if the adjustment option can improve overall results and diminish the non-responder rate.

The Spatz3 Adjustable intragastric balloon (IGB) (Spatz FGIA, Inc. New York, USA) was implanted at the following centers between May and December 2015: University Hospital, Ostrava, Czech Republic, Clinica Opcion Medica, Barcelona, Spain, and Optimal Clinic, Tel Aviv, Israel. Patients were selected according to the well-established criteria for intragastric balloon implantation, consistent with NIH and CE Mark guidelines, and were independently evaluated by members of the staff: gastroenterologists, dieticians, and psychologists. Indications for Spatz3 Adjustable IGB implantation included one of the following: (1) temporary weight loss treatment in a patient with body mass index (BMI) in the range of bariatric surgery (>35) who refuse surgery or are at high risk for surgery, (2) temporary weight loss treatment for a patient without indications for surgery (BMI>29). All patients underwent upper gastrointestinal endoscopy using conscious sedation with or without an anesthetist using one or more of the following medications - Propofol, Midazolam, and Fentanyl.

Balloons were inflated with a mean 464ml (400-500ml) of normal saline with the addition of 2-3 ml of a 1% solution of Methylene Blue (not used in the Czech Republic center). Patients were recovered for 45 minutes and discharged the same day on a once-daily PPI, anti-nausea medications (Aprepitant 125 mg day 1; 80 mg days 2 and 3), ondansetron (8 mg Q6H X 3 days), anti-spasmodic (papaverine 80 mg tid prn), and dietary instructions. After the fifth post-procedure day, a progressive full liquid to soft to solid 1,200-1,400 kcal diet was started. Monthly follow up with dietician and/or doctor (gastroenterologist or endocrinologist) was offered to all patients after implantation. Cognitive behavioral therapy by licensed psychologists was offered in 2 of the 3 centers (206/227 patients) with 6-10 sessions after implantation. Patients who were intolerant to the balloon could be adjusted downward by 100-150 ml. Patients with one or more of the following were offered upward adjustments of the balloon volume (200-400 ml at the discretion of the endoscopist): weight loss plateau; lack of balloon effect; ability to overeat without resultant symptoms (any of the following: nausea, vomiting, bloating, eructation, abdominal pain, acid reflux symptoms). Preparation for an adjustment or extraction procedure required the following diet: 3 days prior- no meat or vegetables; 2 days prior- full liquids; 1 day prior- clear liquids and NPO after midnight. After 12 months of placement, the balloon was deflated by aspiration via standard balloon needle or deflation utilizing the valve, and extraction was completed using a grasping forceps or a polypectomy snare - all under conscious sedation.

ELIGIBILITY:
Inclusion Criteria:

* temporary weight loss treatment in a patient with body mass index (BMI) in the range of bariatric surgery (>35) who refuse surgery or are at high risk for surgery
* temporary weight loss treatment for a patient without indications for surgery (BMI > 29)

Exclusion Criteria:

- none

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a temporary weight loss treatment, with body mass index (BMI) in the range of bariatric surgery (>35) who refuse surgery or are at high risk for surgery or a temporary weight loss treatment without indications for surgery (BMI > 29).
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Weight loss | 8 months
  The achieved weight loss was recorded for the patients in the study.

SECONDARY OUTCOMES:
Balloon intolerance | 8 months
  Intolerance of the intragastric balloon was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Evžen Machytka, MD,PhD, Study Director — University Hospital Ostrava
Locations (4):
- Czechia (2):
  - University of Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
- Optimal Clinic, Tel Aviv, Israel
- Clínica Opcíon Médica, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The authors have no plan make individual participant data available to other researchers.

REFERENCES:
- [Background] Mathus-Vliegen EM. Intragastric balloon treatment for obesity: what does it really offer? Dig Dis. 2008;26(1):40-4. doi: 10.1159/000109385. Epub 2008 Feb 15. PMID 18600014
- [Background] Imaz I, Martinez-Cervell C, Garcia-Alvarez EE, Sendra-Gutierrez JM, Gonzalez-Enriquez J. Safety and effectiveness of the intragastric balloon for obesity. A meta-analysis. Obes Surg. 2008 Jul;18(7):841-6. doi: 10.1007/s11695-007-9331-8. Epub 2008 May 6. PMID 18459025
- [Background] Bonazzi P, Petrelli MD, Lorenzini I, Peruzzi E, Nicolai A, Galeazzi R. Gastric emptying and intragastric balloon in obese patients. Eur Rev Med Pharmacol Sci. 2005 Sep-Oct;9(5 Suppl 1):15-21. PMID 16457125
- [Background] Mion F, Napoleon B, Roman S, Malvoisin E, Trepo F, Pujol B, Lefort C, Bory RM. Effects of intragastric balloon on gastric emptying and plasma ghrelin levels in non-morbid obese patients. Obes Surg. 2005 Apr;15(4):510-6. doi: 10.1381/0960892053723411. PMID 15946431
- [Background] Evans JD, Scott MH. Intragastric balloon in the treatment of patients with morbid obesity. Br J Surg. 2001 Sep;88(9):1245-8. doi: 10.1046/j.0007-1323.2001.01840.x. PMID 11531875
- [Background] Sallet JA, Marchesini JB, Paiva DS, Komoto K, Pizani CE, Ribeiro ML, Miguel P, Ferraz AM, Sallet PC. Brazilian multicenter study of the intragastric balloon. Obes Surg. 2004 Aug;14(7):991-8. doi: 10.1381/0960892041719671. PMID 15329191
- [Background] Genco A, Cipriano M, Bacci V, Cuzzolaro M, Materia A, Raparelli L, Docimo C, Lorenzo M, Basso N. BioEnterics Intragastric Balloon (BIB): a short-term, double-blind, randomised, controlled, crossover study on weight reduction in morbidly obese patients. Int J Obes (Lond). 2006 Jan;30(1):129-33. doi: 10.1038/sj.ijo.0803094. PMID 16189503
- [Background] Doldi SB, Micheletto G, Perrini MN, Rapetti R. Intragastric balloon: another option for treatment of obesity and morbid obesity. Hepatogastroenterology. 2004 Jan-Feb;51(55):294-7. PMID 15025034 (Retraction: PMID 23393648 Hepatogastroenterology. 2012 Nov-Dec;59(120):2683)
- [Background] Roman S, Napoleon B, Mion F, Bory RM, Guyot P, D'Orazio H, Benchetrit S. Intragastric balloon for "non-morbid" obesity: a retrospective evaluation of tolerance and efficacy. Obes Surg. 2004 Apr;14(4):539-44. doi: 10.1381/096089204323013587. PMID 15130235
- [Background] Doldi SB, Micheletto G, Di Prisco F, Zappa MA, Lattuada E, Reitano M. Intragastric balloon in obese patients. Obes Surg. 2000 Dec;10(6):578-81. doi: 10.1381/096089200321594200. PMID 11175969
- [Background] Al-Momen A, El-Mogy I. Intragastric balloon for obesity: a retrospective evaluation of tolerance and efficacy. Obes Surg. 2005 Jan;15(1):101-5. doi: 10.1381/0960892052993558. PMID 15760507
- [Background] Herve J, Wahlen CH, Schaeken A, Dallemagne B, Dewandre JM, Markiewicz S, Monami B, Weerts J, Jehaes C. What becomes of patients one year after the intragastric balloon has been removed? Obes Surg. 2005 Jun-Jul;15(6):864-70. doi: 10.1381/0960892054222894. PMID 15978160
- [Background] Melissas J, Mouzas J, Filis D, Daskalakis M, Matrella E, Papadakis JA, Sevrisarianos N, Charalambides D. The intragastric balloon - smoothing the path to bariatric surgery. Obes Surg. 2006 Jul;16(7):897-902. doi: 10.1381/096089206777822188. PMID 16839490
- [Background] Busetto L, Segato G, De Luca M, Bortolozzi E, MacCari T, Magon A, Inelmen EM, Favretti F, Enzi G. Preoperative weight loss by intragastric balloon in super-obese patients treated with laparoscopic gastric banding: a case-control study. Obes Surg. 2004 May;14(5):671-6. doi: 10.1381/096089204323093471. PMID 15186637
- [Background] Doldi SB, Micheletto G, Perrini MN, Librenti MC, Rella S. Treatment of morbid obesity with intragastric balloon in association with diet. Obes Surg. 2002 Aug;12(4):583-7. doi: 10.1381/096089202762252398. PMID 12194556
- [Background] Totte E, Hendrickx L, Pauwels M, Van Hee R. Weight reduction by means of intragastric device: experience with the bioenterics intragastric balloon. Obes Surg. 2001 Aug;11(4):519-23. doi: 10.1381/096089201321209459. PMID 11501367
- [Background] Courcoulas A, Abu Dayyeh BK, Eaton L, Robinson J, Woodman G, Fusco M, Shayani V, Billy H, Pambianco D, Gostout C. Intragastric balloon as an adjunct to lifestyle intervention: a randomized controlled trial. Int J Obes (Lond). 2017 Mar;41(3):427-433. doi: 10.1038/ijo.2016.229. Epub 2016 Dec 23. PMID 28017964
- [Background] Machytka E, Klvana P, Kornbluth A, Peikin S, Mathus-Vliegen LE, Gostout C, Lopez-Nava G, Shikora S, Brooks J. Adjustable intragastric balloons: a 12-month pilot trial in endoscopic weight loss management. Obes Surg. 2011 Oct;21(10):1499-507. doi: 10.1007/s11695-011-0424-z. PMID 21553304
- [Background] Brooks J, Srivastava ED, Mathus-Vliegen EM. One-year adjustable intragastric balloons: results in 73 consecutive patients in the U.K. Obes Surg. 2014 May;24(5):813-9. doi: 10.1007/s11695-014-1176-3. PMID 24442419
- [Background] Gomez V, Woodman G, Abu Dayyeh BK. Delayed gastric emptying as a proposed mechanism of action during intragastric balloon therapy: Results of a prospective study. Obesity (Silver Spring). 2016 Sep;24(9):1849-53. doi: 10.1002/oby.21555. Epub 2016 Jul 28. PMID 27465076
- [Background] Mathus-Vliegen EM, Tytgat GN. Intragastric balloon for treatment-resistant obesity: safety, tolerance, and efficacy of 1-year balloon treatment followed by a 1-year balloon-free follow-up. Gastrointest Endosc. 2005 Jan;61(1):19-27. doi: 10.1016/s0016-5107(04)02406-x. PMID 15672051
- [Background] Dastis NS, Francois E, Deviere J, Hittelet A, Ilah Mehdi A, Barea M, Dumonceau JM. Intragastric balloon for weight loss: results in 100 individuals followed for at least 2.5 years. Endoscopy. 2009 Jul;41(7):575-80. doi: 10.1055/s-0029-1214826. Epub 2009 Jul 8. PMID 19588283
- [Background] Al Kahtani K, Khan MQ, Helmy A, Al Ashgar H, Rezeig M, Al Quaiz M, Kagevi I, Al Sofayan M, Al Fadda M. Bio-enteric intragastric balloon in obese patients: a retrospective analysis of King Faisal Specialist Hospital experience. Obes Surg. 2010 Sep;20(9):1219-26. doi: 10.1007/s11695-008-9654-0. Epub 2008 Aug 28. PMID 18752030